CLINICAL TRIAL: NCT05201911
Title: A Single Arm, Single Dose Study to Characterize the Biodistribution of 124I-Labeled AT-03 in Select Organs in Patients With Systemic Amyloidosis
Brief Title: A Study to Characterize the Biodistribution of 124I-Labeled AT-03 in Patients With Systemic Amyloidosis
Acronym: AT03-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Attralus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AT03-001
Record Dates: First submitted 2021-12-02; First posted 2022-01-21 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Amyloidosis; Systemic
Keywords: Amyloid Light-Chain (AL); Transthyretin Amyloidosis (ATTR); Leukocyte chemotactic factor 2 amyloidosis (ALECT2); All other forms of systemic amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Injection of I-124 AT03. (Experimental): Single arm only, no placebo or comparator
  Interventions: Drug: 124I-AT03

INTERVENTIONS:
Drug: 124I-AT03 — IV injection of the radiolabeled compound on day 1 followed by Positron Emission Tomography/Computed Tomography (PET/CT) scanning on Days 2, 4 and 8 to. The first 3 subjects enrolled will have two additional scans on Day 1.

SUMMARY:
This is a single center Phase 1 study is to evaluate the biodistribution of radiolabeled AT-03 in patients with systemic amyloidosis.

DETAILED DESCRIPTION:
Eligible subjects will receive a single dose of radiolabeled AT-03, a fusion protein of serum amyloid P and a single chain Fc receptor. Repeat Positron Emission Tomography/Computed Tomography (PET/CT) scans will be performed over a ~7 day period to assess the biodistribution of AT-03 to amyloid-containing tissues in patients with systemic amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Understands the study procedures and capable of giving signed informed consent, as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Male or female ≥18 years of age.
3. Has a confirmed diagnosis of Amyloid Light-Chain (AL), Transthyretin Amyloidosis (ATTR), or Leukocyte chemotactic factor 2 amyloidosi (ALECT2), or any other forms of systemic amyloidosis based on any one of the following:

   1. a histologic confirmation with a biopsy containing deposits of apple-green birefringent, congophilic material;
   2. genetic screening with presence of amyloid-related pathology; and/or
   3. amyloid-specific imaging study.
4. Has known involvement of at least one thoracoabdominal organ (excluding peripheral nervous system) by clinical history (e.g., imaging consistent with amyloid deposition, organ biopsy, elevated amyloid-related biomarkers, etc.).
5. For women of childbearing potential: agreement to remain as abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 90 days after the last dose of study intervention.

   1. A woman is considered of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
   2. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices.
   3. Contraception methods that do not result in a failure rate of <1% per year such as cap, diaphragm, or sponge with spermicide, or male or female condom with or without spermicide, are not acceptable.
   4. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
6. For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm, as defined below:

   1. With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 30 days plus 90 days (a spermatogenesis cycle) after the last dose of study intervention. Men must refrain from donating sperm during this same time period.

Exclusion Criteria:

1. Is pregnant or breast-feeding.
2. Is mentally or legally incapacitated, has significant emotional problems at the time of the study, or has a history of psychosis.
3. Has participated in another nuclear medicine amyloid imaging clinical trial protocol and received tracer injection in the 4 months prior to Screening.
4. Has a significant co-morbidity (e.g., ECOG score of 3 or greater), NYHA Class IV heart failure, uncontrolled infection, or other ongoing serious illness.
5. Has a known allergy to iOSAT iodine treatment.
6. Has end-stage renal disease and is receiving hemodialysis or peritoneal dialysis.
7. Has received an investigational agent within five half-lives of the agent or 30 days, whichever is longer, prior to Screening.
8. Has any illness that, in the opinion of the Investigator, might confound the results of the study or pose additional risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
To measure the tissue distribution of 124I-AT-03 in select organs in patients with systemic amyloidosis as shown in the Positron Emission Tomography/Computed Tomography (PET/CT scans) series. | Day 4.
  Visual determination of 124I-AT-03 uptake in the heart, kidneys, liver and spleen (positive or negative) at Days 4 and 6.
To measure the tissue distribution of 124I-AT-03 in select organs in patients with systemic amyloidosis as shown in the Positron Emission Tomography/Computed Tomography (PET/CT scans) series. | Day 6.
  Visual determination of 124I-AT-03 uptake in the heart, kidneys, liver and spleen (positive or negative) at Days 4 and 6.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events. | Assessed from time of consent through the day 28 follow-up phone call.
  Incidence of treatment-emergent adverse events from Day 1 to Day 28.
Number of participants with abnormal laboratory test results. | Assessed from time of consent through Day 6.
  Change from Baseline in clinical laboratory values at Days 4 and 6.
Whole blood radioactivity of 124I-AT-03 in subjects with systemic amyloidosis. | Days 1, 4, and 6.
  Whole body radiation dose by dosimetry in all enrolled subjects. Whole blood radioactivity (corrected for radioactive decay).
Selected tissue-bound half-life of 124I-AT-03 in subjects with systemic amyloidosis. | Days 4 and 6.
  Organ specific radioactivity for the heart, kidneys, liver, and spleen at Days 4 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bell, MD, Study Director — Attralus, Inc.
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No